CLINICAL TRIAL: NCT03991364
Title: Comparison of Robot-assisted Gait Training According to Gait Speed in Participants With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2019-01-002
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: Robot-assisted gait training; stroke; gait speed
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constant gait speed group (Experimental): experimental group that applied the speed of the robot-assisted gait training constantly
  Interventions: Other: Constant gait speed group
- Increasing gait speed group (Other): control group that applied the gradual increase of the speed of the robot-assisted gait training
  Interventions: Other: Increasing gait speed group

INTERVENTIONS:
Other: Constant gait speed group — The speed of the robot-assisted gait treatment is constantly applied for 5 times a week for 2 weeks.
  Arms: Constant gait speed group
Other: Increasing gait speed group — The speed of the robot-assisted gait treatment is gradually increase for 5 times a week for 2 weeks.
  Arms: Increasing gait speed group

SUMMARY:
Comparison of the experimental group that applied the speed of the robot-assisted gait training constantly and the control group that applied the gradual increase of the speed of the robot-assisted gait training.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Functional ambulation category score ≥ 3

Exclusion Criteria:

* History of surgery of affected lower limb
* Fracture of affected lower limb

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure (EE) | 2 weeks after baseline
  EE(kcal/min): energy expenditure per minute

SECONDARY OUTCOMES:
Energy expenditure (EE) | baseline, 1 weeks after baseline, 3 weeks after baseline
  EE(kcal/min): energy expenditure per minute
Heart rate (HR) | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  Cardiac frequency
Volume of Oxygen (VO2) | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  O2 consumption/1min
Respiratory Quotient (R) | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  Respiratory quotient
Metabolic equivalent (METS) | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min
oxygenated hemoglobin (OxyHb) | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  oxygenated hemoglobin concentration of cortical activation
deoxygenated hemoglobin (DeoxyHb) | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  deoxygenated hemoglobin concentration of cortical activation
Lower extremity Fugl-Meyer Assessment | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  Fugl-Meyer Assessment uses to examine the motor function and coordination of affected lower extremity. It includes 17 items of a 3-point ordinal scale, ranging 0-34, with higher scores indicating lower impairment.
Functional Ambulation Category | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  Functional Ambulation Category is used to assess gait ability with 6 levels ranging from 0 to 5 on the basis of the amount of physical support required, regardless of use of an assistive device
10m walk test | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  10m walk test is used to examine gait speed, in which participant was asked to walk on a 14 meter of walkway wearing harness with two conditions; with the fastest speed or with self-selected comfortable speed.
timed up and go test | baseline, 1 weeks after baseline, 2 weeks after baseline, 3 weeks after baseline
  simple test used to assess a person's mobility and requires both static and dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea